CLINICAL TRIAL: NCT02623114
Title: Comprehensive Pathophysiological Study Based on the Core Neurocognitive Deficits and Development of Biological Markers of Treatment Response in Attention Deficit Hyperactivity Disorder
Brief Title: Attention-deficit/Hyperactivity Disorder Translational Center for Identifying Biomarkers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Childrens Hospital (Other)
Responsible Party: Principal Investigator, Booog Nyung Kim, Professor, Seoul National University Childrens Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0720151002
Record Dates: First submitted 2015-11-29; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): ADHD patients with methylphenidate administration Generic names include concerta, metadata and penid. The initial dosage was fixed for 2 weeks and then adjusted according to the clinician's judgement. The patients visited the hospital at week 2,4,6,8,16,24, 9months, 12,15,18,21,24 months.
  Interventions: Drug: methylphenidate
- Atomoxetine (Experimental): ADHD patients with atomoxetine administration Generic names include strattera. The initial dosage was fixed for 2 weeks and then adjusted according to the clinician's judgement. The patients visited the hospital at week 2,4,6,8,16,24, 9months, 12,15,18,21,24 months.
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: methylphenidate — The patients received a fixed dose of medication for 2 weeks. The dose was increased according to the clinician's judgment. The patients came to the hospital at week 2,4,6,8,16,24wks, 9, 12,15,18,21,24 months
  Other Names: concerta, metadate, penid
  Arms: Methylphenidate
Drug: atomoxetine — The patients received a fixed dose of medication for 2 weeks. The dose was increased according to the clinician's judgment. The patients came to the hospital at week 2,4,6,8,16,24wks, 9, 12,15,18,21,24 months
  Other Names: strattera
  Arms: Atomoxetine

SUMMARY:
The purpose of this study was to identify genetic, brain morphologic, and environmental biomarkers that contribute to the pathophysiology of attention-deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The investigators planned to recruit ADHD and healthy controls from the age of 6 to 17.

Genetic data including dopamine, norepinephrine, serotonin, neurotropic factors, glutamate-related genes will be genotyped.

Environmental disruptors including phthalate and cotinine will be analyzed. Brain MRI data including T1, diffusion tensor imaging (DTI), resting state functional MRI (rsfMRI) will be obtained.

Neuropsychological tests including continuous performance test, Stroop test, Children's color trail test, Wisconsin card sorting test will be conducted.

The investigators plan to identify biomarkers of ADHD using an integrative approach of genetic, environmental, neuroimaging and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of attention-deficit/hyperactivity disorder confirmed using the Kiddie-Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version- Korean Version (K-SADS-PL-K).
* IQ over 70

Exclusion Criteria:

* Intelligence quotient (IQ) < 70
* A hereditary genetic disorder
* A current/past history of brain trauma, organic brain disorder, seizure, or any neurological disorder
* Autism spectrum disorder, communication disorder, or learning disorder
* Schizophrenia or any other childhood-onset psychotic disorder
* Major depressive disorder or bipolar disorder
* Tourette's syndrome or chronic motor/vocal tic disorder
* obsessive-compulsive disorder
* A history of methylphenidate treatment lasting more than 1 year or received within the previous 4 weeks

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-08 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Treatment response measured by decrease in ADHD-RS scale | 6 months
  Changes in the Parent rated ADHD-Rating Scale - IV (ADHD-RS), which is an 18 item scale, with 9 items assessing inattention and 9 items assessing hyperactivity/impulsivity. It is the most widely used scale to measure symptom severity of attention-deficit/hyperactivity disorder.
Treatment response measured by CGI-I score | 6 months
  The Clinical Global Impression - Improvement (CGI-I) scale is a clinician rated scale used to measure improvement in symptoms. It ranges from 1 to 7, with 1 meaning very much improved, and 7 meaning very much worse.
Treatment response measured by changes in CPT score | 6 months
  The continuous performance test (CPT) is an objective measurement of ADHD symptom severity. It is a computerized test and the results are presented in 4 variables : omission errors, commission errors, response time, response time variability.

SECONDARY OUTCOMES:
Treatment response measured by decrease in ADHD-RS scale | 1 year
  The ADHD-RS scale is described in primary outcome measures.
Side effects measured using the side effect rating scale (SRS) | 1 year
  The side effect rating scale (SRS) is a parent rated scale, measuring side effects of multiple domains in the previous 2 week period.
Treatment response measured by CGI-I score | 1 year
  The CGI-I scale is described in primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Boong-nyun Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea